CLINICAL TRIAL: NCT00573378
Title: A Combination of Imatinib or Nilotinib Together With Pegylated Interferon-α2b in Chronic-Phase Chronic Myeloid Leukemia: A Phase II Pilot Study Targeting Both the Primitive and Differentiated CML Progenitor Populations
Brief Title: Imatinib or Nilotinib With Pegylated Interferon-α2b in Chronic Myeloid Leukemia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2006.128; HUM9600 (Other: University of Michigan Medical IRB)
Record Dates: First submitted 2007-12-13; First posted 2007-12-14 (Estimated); Results first posted 2023-01-25 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Chronic Myeloid Leukemia
Keywords: CML
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — peginterferon alfa-2b

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- PEG-IFN-a2b (Experimental)
  Interventions: Drug: PEG-IFN-a2b

INTERVENTIONS:
Drug: PEG-IFN-a2b — Patients will receive pegylated interferon α-2b (Pegintron®) (PEG-IFN-α2b) 150 µg subcutaneously, once a week. Patients and/or caregivers identified by the patient will be taught how to perform subcutaneous injections of the PEG-IFN-α2b by trained nurses in the chemotherapy infusion center at the University of Michigan Comprehensive Cancer Center. Those patients who do not feel comfortable receiving the injections outside of the cancer center, or are deemed unreliable in administering injections per the training nurse, will return to the cancer center infusion room on a weekly basis to receive subsequent injections.
  Other Names: Pegintron®

SUMMARY:
To investigate whether patients with chronic-phase chronic myeloid leukemia (CP-CML) who have achieved a complete cytogenetic response (CCyR) on imatinib (IM) or nilotinib (N) can then be treated with a combination of the tyrosine kinase inhibitor (TKI) and interferon-α2b (PEG-IFN-a2b, [IFN]) for 2 years, subsequently have their therapy discontinued, and then maintain a durable molecular response off all therapy. Relapse-free survival (RFS) rate 1 year after discontinuation of the TKI and IFN will be the measurement of this objective.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a diagnosis of Philadelphia chromosome positive (Ph+) chronic myeloid leukemia in chronic phase by having met all of the following criteria at the time of their initial diagnosis:
* Cytogenetic confirmation of Philadelphia chromosome or variants of the t(9;22) translocations. Patients may have secondary chromosomal abnormalities in addition to the Philadelphia chromosome.
* Peripheral blood or bone marrow blast count < 10%.
* Peripheral blood basophil count < 20%.
* Platelet count ≥ 100,000 x 109/L.
* If the peripheral blood counts are unavailable from the time of their original diagnosis, but there is no evidence of accelerated- or blast-phase disease from prior clinical or other medical records, then they will be allowed to participate.
* Patients must be eighteen years of age or older.
* Patients must be actively receiving treatment for their CML with a a tyrosine kinase inhibitor, either imatinib or nilotinib.
* Patients may be receiving imatinib mesylate. Patients must be on imatinib mesylate for a minimum of 2 years, and be on a stable dose for at least one consecutive year leading up to enrollment.
* Patients may be receiving nilotinib (Tasigna) as frontline therapy or as second line therapy if the reason for the switch from imatinib to nilotinib was intolerance to imatinib. Patients cannot have been switched from imatinib to nilotinib because of a concern or demonstration for resistance to frontline imatinib. Patients must be on nilotinib for a minimum of 2 years, and be on a stable does for at least one consecutive year leading up to enrollment.
* Patients must have an ongoing complete hematologic response (CHR) on a a TKI (imatinib or nilotinib), defined as follows:
* WBC ≤ 10 x 109/L.
* Platelet count < 450,000 x 109/L.
* No blasts or promyelocytes in peripheral blood.
* No evidence of disease-related symptoms and extramedullary disease, including the liver and spleen.
* Patients must have a complete cytogenetic response (CCyR) on a TKI (imatinib or nilotinib) for a minimum of 1 year leading up to enrollment. Complete cytogenetic response is defined as 0% Ph+ cells in metaphase, in the bone marrow and/or a negative peripheral blood FISH analysis for the Bcr-Abl gene fusion, and an ongoing CCyR must be confirmed by bone marrow aspirate cytogenetics and/or peripheral blood FISH for Bcr-Abl within 4 weeks of starting treatment.
* Patients may have a negative quantitative RT-PCR (qPCR) for BCR-ABL at the time of enrollment, but if the qPCR is positive, patients cannot have greater than 1% bcr-ABl / Abl /ABL transcript, present in 2 consecutive qPCR analyses, performed at least 3 months apart, in the 6 to 12 months leading up to enrollment.
* Patients must have an ECOG performance status of 0-2 (Appendix 13.1).
* All patients must be informed of the investigational nature of this study and standard alternative therapy. All patients must sign and give written informed consent in accordance with institutional and federal guidelines.

Exclusion Criteria:

* Patients who have had prior progression of their CML to accelerated phase or blast crisis.
* Patients who have previously undergone hematopoietic stem cell transplantation.
* Patients who have previously been treated with interferon-α.
* Patients with an absolute neutrophil count (ANC) < 1500/mm3 and/or a platelet count < 100,000/mm3.
* Patients with serum bilirubin, SGOT[AST], SGPT[ALT], or serum creatinine > 1.5 x the upper limit of normal (ULN).
* Patients with an INR or PTT > 1.5 x ULN, with the exception of patients on treatment with oral anticoagulants.
* Patients with uncontrolled medical diseases such as diabetes mellitus, neuropsychiatric disorders, infection, angina, severe hypertension, pulmonary disease (chronic obstructive pulmonary disease [COPD] with hypoxemia), major organ malfunction (liver, kidney) or class III or IV cardiac disease as defined by the New York Heart Association Criteria.
* Patients who are (a) pregnant, (b) breast feeding, (c) of childbearing potential without a negative pregnancy test prior to Study Day 1, and (d) male or female of childbearing potential unwilling to use barrier contraceptive precautions throughout the trial (postmenopausal women must be amenorrheic for at least 12 months to be considered of non-childbearing potential).
* Patients with a history of another active malignancy within the last five years, which required treatment with chemotherapy, hormonal therapy, or radiation therapy. Exceptions to this rule include basal cell and squamous cell skin carcinomas or cervical carcinoma in situ.
* Patients with a history of non-compliance to medical regimens or who are considered potentially unreliable.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2007-09 (Actual); Primary Completion 2010-10 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dale L. Bixby, M.D., Principal Investigator — University of Michigan
Locations (1):
- Universtiy of Michigan, Ann Arbor, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- PEG-IFN-a2b: PEG-IFN-a2b: Patients receive pegylated interferon α-2b (Pegintron®) (PEG-IFN-α2b) 150 µg subcutaneously, once a week.
Period: Overall Study
Arm/Group | PEG-IFN-a2b
Started | 12
Evaluable for Primary Outcome Measure | 1
Completed | 0
Not Completed | 12

BASELINE CHARACTERISTICS:
Arm/Group | PEG-IFN-a2b
Number analyzed (Participants) | 12
Age, Continuous [Mean (Full Range); unit: years] | 39 [19 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 11
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Relapse-free Survival (RFS) Rate 1 Year After Discontinuation of the TKI and IFN
Description: To investigate whether patients with chronic-phase chronic myeloid leukemia (CP-CML) who have achieved a complete cytogenetic response (CCyR) on imatinib (IM) or nilotinib (N) can then be treated with a combination of the tyrosine kinase inhibitor (TKI) and interferon-α2b (PEG-IFN-a2b, [IFN]) for 2 years, subsequently have their therapy discontinued, and then maintain a durable molecular response off all therapy. Relapse-free survival (RFS) rate 1 year after discontinuation of the TKI and IFN will be the measurement of this objective.
Time Frame: 3 years (2 years of treatment with TKI and IFN + 1 year of follow-up)
Measure: Count of Participants; unit: Participants
Arm/Group | PEG-IFN-a2b
Number analyzed (Participants) | 1
Participants | 0

2. Secondary Outcome: Quantitative Reverse Transcriptase-polymerase Chain Reaction (qRT-PCR) for the Bcr-Abl Transcript.
Description: To determine whether the addition of PEG-IFN-a2b to a TKI (imatinib or nilotinib) improves upon the quality of the molecular remission seen with TKI alone, as measured by quantitative reverse transcriptase-polymerase chain reaction (qRT-PCR) for the Bcr-Abl transcript.
Time Frame: 3 years (2 years of treatment with TKI and IFN + 1 year of follow-up)
Population: Because there were no molecular remissions at 1 year post treatment discontinuation (measure #1), there was no basis for this analysis. There is no data to summarize.
Arm/Group | PEG-IFN-a2b
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Throughout study treatment and for 30 days post discontinuation of study treatment (25 months). Patients will continue in follow up; however, AEs will no longer be collected.
Description: Grade 3 and/or 4 serious adverse events (SAE) that are unexpected and definitely, probably or possibly related to protocol therapy are reported.
Arm/Group | PEG-IFN-a2b
All-Cause Mortality (participants affected / at risk) | 1/12
Serious Adverse Events (participants affected / at risk) | 1/12
Other Adverse Events (participants affected / at risk) | 0/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PEG-IFN-a2b (N=12)
Urethral obstruction (Renal and urinary disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes